CLINICAL TRIAL: NCT06149299
Title: Comparison of Pain Relief and Block Success of Great Occipital Nerve Block Using Different Approach Method at C2 Level
Brief Title: Great Occipital Nerve Block Using Different Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-10-025
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interfascial plane group (Placebo Comparator): injection into inferfascial plane
  Interventions: Procedure: Greater occipital nerve block
- intramuscular group (Experimental): injection into obliqus capitis inferior muscle
  Interventions: Procedure: Greater occipital nerve block

INTERVENTIONS:
Procedure: Greater occipital nerve block — Greater occipital nerve block using ultrasound guidance

SUMMARY:
Great occipital nerve (GON) block is commonly applied for the pain management of occipital neuralgia, migraine, and cervicogenic headache. The GON orginates from the medial branch of the dorsal ramus of the C2 spinal nerve with variable contribution from the C3 dorsal ramus. After emerging from the suboccipital triangle, the nerve courses cephalad in an oblique trajectory between the semispinalis capitis (SC) and obliqus capitis inferior (OCI) muscles. This area was recognized as a potential location for GON injury. The nerve then passes through the trapezius muscle and courses medial to the occipital artery as it ascends to innervate the posterior scalp.

Many practitioners perform GON injections using a conventional approach, relying solely on superficial bone-based anatomic landmarks to infiltrate local anesthetic and corticosteroid around the nerve at the level of the superior nuchal line.

Some clinicians also use fluoroscopy to confirm the location of bony landmarks. The ambiguity of these injections poses a risk of anesthetizing adjacent structures or injecting into vessels, such as the occipital artery. Very limited research has been done to quantify the risk of these injections, but a complication rate of 5% to 10% has been reported, including headache, dizziness, blurred vision, and syncope.

Ultrasound guidance is increasingly used to mitigate these risks and improve the efficacy of GON injections. Multiple studies have demonstrated successful ultrasound-guided GON blockade at the superior nuchal line and improvement in pain scores compared with nonguided injections.

C2 level GON block using ultrasound targets interfascial plane between OCI and SC muscles. However, a pain physician who begins ultrasound guided injections migth feel very difficult targeting interfascial plane exactly.

Since GON orginiates from deep space of suboccipital triangle, it is expected that injection within OCI muscle might have similar effect with the effect of injection into interfascial plane.

We assume that if the local anesthetics is injected within OCI muscle, the effect of GON block will be generated by the diffusion of injected local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Cervicogenic headache
* Migraine
* Occipital neuralgia

Exclusion Criteria:

* bilateral headache
* cervical spine surgery within 1 year before
* loss of sensory sensation at the dermatome of GON innervation
* anatomical defect at the region of procedure
* coagulopathy
* pregnancy or breast feeding
* allergy to local anesthetics

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale | Baseline, 30 minutes, 2 weeks, 4 weeks after the completion of GON block
  Numerical rating scale after GON block
block success | Baseline, 30 minutes after the completion of GON block
  block success after GON block

SECONDARY OUTCOMES:
Side effect after GON block | Baseline, 30 minutes after the completion of GON block
  Side effect after GON block

CONTACTS AND LOCATIONS:
Locations (1):
- Hong ji HEE, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No